CLINICAL TRIAL: NCT00083694
Title: UARK, 98-032, Thalidomide Anti-Angiogenesis Therapy of Relapsed or Refractory Leukemia
Brief Title: Thalidomide Anti-Angiogenesis Therapy of Relapsed or Refractory Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Celgene Corporation (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UARK 98-032
Record Dates: First submitted 2004-05-27; First posted 2004-05-31 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2010-07

CONDITIONS: Leukemia
Keywords: Leukemia; Thalidomide; relapsed
MeSH Terms: conditions — Leukemia; Recurrence | interventions — Thalidomide

INTERVENTIONS:
Drug: Thalidomide

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Thalidomide in patients with leukemia.

DETAILED DESCRIPTION:
Patients will take Thalidomide tablets at bedtime daily until remission. The dose will be increased gradually and modified according to side-effects. The drug will be given daily up to the time of complete remission then as long as it is beneficial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of refractory or relapsed leukemia: acute leukemia, CML, CLLm and MDS.
* Signed informed consent, including patient agreeing to use safe contraceptive methods during the treatment and for at least 4 months after the treatment is completed
* Serum creatinine < or = 2.5mg/dL
* Serum bilirubin< or = 2.5mg/dL
* Negative pregnancy test
* Age 18 years or older
* Performance status < or = 3

Exclusion Criteria:

* Pregnant or lactating women
* Concurrent treatment with cytotoxic chemotherapy, or radiation
* History of seizures, neurotoxicity, or active CNS disease
* Serious infections not controlled by antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 1998-08; Study Completion 2005-05

PRIMARY OUTCOMES:
To evaluate the efficacy and safety of Thalidomide in patients with leukemia.

CONTACTS AND LOCATIONS:
Overall Officials: Barthel Barlogie, M.D., Ph.D., Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences/MIRT, Little Rock, Arkansas, United States

REFERENCES:
- See also: Myeloma Institute for Research & Therapy website — http://myeloma.uams.edu